CLINICAL TRIAL: NCT02446418
Title: A 6-month, Open Label, Randomised, Efficacy Study to Evaluate Fluticasone Furoate (FF, GW685698)/Vilanterol (VI, GW642444) Inhalation Powder Delivered Once Daily Via the Dry Powder Inhaler ELLIPTA™ Compared With Usual ICS/LABA Maintenance Therapy Delivered by Dry Powder Inhaler in Subjects With Persistent Asthma
Brief Title: A Study to Compare the Efficacy of Fluticasone Furoate/Vilanterol Inhalation Powder With Usual Inhaled Corticosteroids (ICS)/Long Acting Beta Agonists (LABA) in Persistent Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 116492
Record Dates: First submitted 2015-05-14; First posted 2015-05-18 (Estimated); Results first posted 2019-01-14 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2018-06

CONDITIONS: Asthma
Keywords: dry powder inahler; vilanerol; efficacy; safety; fluticasone furoate; quality of life
MeSH Terms: conditions — Asthma | interventions — fluticasone furoate; vilanterol; Fluticasone; Salmeterol Xinafoate; Budesonide; Formoterol Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluticasone Furoate/Vilanterol (Experimental): Subjects will receive FF/VI 92 micrograms (mcg)/22 mcg or FF/VI 184 mcg/22 mcg as decided by the investigator QD via ELLIPTA DPI for 24 weeks.
  Interventions: Drug: Fluticasone Furoate; Drug: Vilanterol
- FP/S OR BUD/F (Active Comparator): Subjects will receive FP/S (250 mcg/50 mcg or 500 mcg/50mcg) twice daily via DISKUS or BUD /F (200 mcg/6mcg or 400 mcg/12mcg one or two inhalations) twice daily via TURBUHALER DPI as decided by the investigator for 24 weeks.
  Interventions: Drug: Fluticasone propionate; Drug: Salmeterol; Drug: Budesonide; Drug: Formoterol Fumarate

INTERVENTIONS:
Drug: Fluticasone Furoate — FF 92 mcg or 184 mcg blended with lactose administered once daily via ELLIPTA DPI
  Arms: Fluticasone Furoate/Vilanterol
Drug: Vilanterol — Vilanterol 22 mcg blended with lactose and magnesium stearate administered once daily via ELLIPTA DPI
  Arms: Fluticasone Furoate/Vilanterol
Drug: Fluticasone propionate — FP 250 mcg or 500 mcg blended with lactose administered twice daily via DISKUS DPI
  Arms: FP/S OR BUD/F
Drug: Salmeterol — Salmeterol 50 mcg blended with lactose administered twice daily via DISKUS DPI
  Arms: FP/S OR BUD/F
Drug: Budesonide — Budesonide 200 mcg or 400 mcg blended with lactose administered twice daily via TURBUHALER DPI
  Arms: FP/S OR BUD/F
Drug: Formoterol Fumarate — Formoterol Furoate 6 mcg or 12 mcg blended with lactose administered twice daily via TURBUHALER DPI
  Arms: FP/S OR BUD/F

SUMMARY:
The combination of FF, an ICS and VI, an orally inhaled LABA has been developed as a once-daily combination therapy for the long-term maintenance treatment of asthma in adults and children >=12 years of age. Pivotal phase III studies have demonstrated the safety and efficacy of FF/VI in asthma. However, it is increasingly acknowledged that randomised clinical trials tend to be highly controlled and enrol a more highly selected subject population than is expected to be prescribed the medication post-approval. There is a need for data in a more representative population in close to a 'real life' conditions, where physicians have the ability to choose the best treatment in their view for any individual subject and adapt treatments to subjects' characteristics and response. This multi-center, open-label, randomized, parallel group study will evaluate the efficacy and safety of FF/VI compared with two usual ICS/LABA fixed combination (fluticasone propionate/salmeterol [FP/S] or budesonide/formoterol [BUD/F]) in subjects with persistent asthma, in a "close to real life" settings. FF/VI will be administered once-daily (QD) via ELLIPTA dry powder inhaler (DPI) and FP/S or BUD/F will be administered twice daily (BID) via DISKUS™ and TURBUHALER™ DPI respectively. ELLIPTA is a new powder inhaler designed to be easy to use. The total duration of subject participation will be approximately 6 months (24 weeks). ELLIPTA and DISKUS are registered trademarks of the GSK group of companies. TURBUHALER is a registered trademark of AstraZeneca.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent: Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in this protocol.
* Gender and Age: Male or female subjects aged >=18 and <=75years of age at Screening visit.

Female subject is eligible to participate if she is not pregnant (as confirmed by a negative urine human chorionic gonadotrophin [hCG] test), not lactating, and at least one of the following conditions applies:

Non-reproductive potential defined as: Pre-menopausal females with one of the following - Documented tubal ligation; Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion; Hysterectomy; Documented Bilateral Oophorectomy. Postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone [FSH] and estradiol levels consistent with menopause [refer to laboratory reference ranges for confirmatory levels]); Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.

Reproductive potential and agrees to follow one of the options listed below in the GSK Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) requirements from 30 days prior to the first dose of study medication and until Week 24.

GSK Modified List of Highly Effective Methods for Avoiding Pregnancy in FRP:

This list does not apply to FRP with same sex partners, when this is their preferred and usual lifestyle or for subjects who are and will continue to be abstinent from penile-vaginal intercourse on a long term and persistent basis: Contraceptive subdermal implant that meets the Standard Operating Procedure (SOP) effectiveness criteria including a <1percent rate of failure per year, as stated in the product label; Intrauterine device or intrauterine system that meets the SOP effectiveness criteria including a <1 percent rate of failure per year, as stated in the product label; Oral Contraceptive, either combined or progestogen alone; Injectable progestogen; Contraceptive vaginal ring; Percutaneous contraceptive patches; Male partner sterilization with documentation of azoospermia prior to the female subject's entry into the study, and this male is the sole partner for that subject; Male condom combined with a vaginal spermicide (foam, gel, film, cream, or suppository); These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.

* Type of subject: Subjects with documented physician's diagnosis of asthma >=1 year, unsatisfactorily controlled asthma (ACT <20 at Screening and Randomisation visit) treated by ICS alone and intended to be treated by ICS/LABA maintenance therapy; France Only: A subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a Social Security category.
* Current Asthma Therapy: All subjects must be prescribed maintenance therapy and receiving ICS alone without LABA for at least 4 weeks prior to Randomisation visit; Other background asthma medication such as anti-leukotrienes or theophylline is permitted as an alternative to ICS alone, if initiated at least 4 weeks prior to screening visit.
* Subject questionnaires Subjects must be able to complete the questionnaires themselves.

Exclusion Criteria:

* History of Life-threatening asthma: Defined for this protocol as an asthma episode that required intubation and/or was associated with hypercapnea, respiratory arrest or hypoxic seizures within the last 6 months before Screening and Randomisation visit.
* Subjects having a severe and unstable asthma, with ACT score < 15 at Visit 1 and at Visit 2, and/or a history of repeated severe exacerbations (3/year) and/or a severe exacerbation in the previous 6 weeks before Visit 1 and Visit 2.
* Chronic obstructive pulmonary disease (COPD) Respiratory Disease: A subject must not have current evidence or diagnosis of chronic obstructive pulmonary disease at Screening visit.
* Current or former cigarette smokers with a history of cigarette smoking of >=10 pack-years at screening [number of pack years = (number of cigarettes per day / 20) x number of years smoked (e.g., 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years)].
* Other diseases/abnormalities: Subjects with historical or current evidence of uncontrolled or clinically significant disease at Screening and Randomisation visit. Significant is defined as any disease that, in the opinion of the Investigator, would put the safety of the subject at risk through participation, or which would affect the efficacy or safety analysis if the disease/condition exacerbated during the study.
* Subjects with a history of adverse reaction including immediate or delayed hypersensitivity to any intranasal, inhaled, or systemic corticosteroid and LABA therapy and to components of the inhalation powder (e.g., lactose, magnesium stearate) at Screening and Randomisation visit. In addition, subjects with a history of severe milk protein allergy that, in the opinion of the Investigator, contraindicates the subject's participation will also be excluded.
* Investigational Medications: A subject must not have used any investigational drug within 30 days prior to Randomisation visit or within five half-lives (t½) of the prior investigational study (whichever is longer of the two), (if unsure discuss with the medical monitor prior to screening).
* Chronic user of systemic corticosteroids: A subject who, in the opinion of the Investigator, is considered to be a chronic user of systemic corticosteroids for respiratory or other indications (if unsure discuss with the medical monitor prior to screening) at Screening visit.
* Subjects treated by the monoclonal antibody omalizumab or mepolizumab at Visit 1. Treatment with omalizumab or mepolizumab is not allowed during the study.
* Subjects involved in other clinical trials at Screening visit.
* Affiliation with Investigator Site: Is an investigator, sub-investigator, study coordinator, employee of a participating investigator or study site, or immediate family member of the aforementioned that is involved in this study.
* Subjects who plan to move away from the geographical area where the study is being conducted during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 423 (Actual)
Dates: Start 2015-07-09 (Actual); Primary Completion 2017-07-20 (Actual); Study Completion 2017-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (81):
- France (68):
  - GSK Investigational Site, Amiens
  - GSK Investigational Site, Angers
  - GSK Investigational Site, Avelin
  - GSK Investigational Site, Bassussarry
  - GSK Investigational Site, Beauzelle
  - GSK Investigational Site, Bersée
  - GSK Investigational Site, Bécon-les-Granits
  - GSK Investigational Site, Béziers
  - GSK Investigational Site, Biarritz
  - GSK Investigational Site, Bourg-des-Comptes
  - GSK Investigational Site, Broglie
  - GSK Investigational Site, Bruay-la-Buissière
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Cannes
  - GSK Investigational Site, Carbon-Blanc
  - GSK Investigational Site, Châtellerault
  - GSK Investigational Site, Colombey-les-Belles
  - GSK Investigational Site, Coulounieix-Chamiers
  - GSK Investigational Site, Cournonterral
  - GSK Investigational Site, Dessenheim
  - GSK Investigational Site, Dijon
  - GSK Investigational Site, Dinard
  - GSK Investigational Site, Donges
  - GSK Investigational Site, Ermont
  - GSK Investigational Site, Fléville-devant-Nancy
  - GSK Investigational Site, Gémenos
  - GSK Investigational Site, Gondreville
  - GSK Investigational Site, Grenay
  - GSK Investigational Site, Guesnain
  - GSK Investigational Site, Hatten
  - GSK Investigational Site, Hinx
  - GSK Investigational Site, La Bouëxière
  - GSK Investigational Site, La Fôret Sur Sèvres
  - GSK Investigational Site, La Riche
  - GSK Investigational Site, Lambersart
  - GSK Investigational Site, Laval
  - GSK Investigational Site, Le Blanc-Mesnil
  - GSK Investigational Site, Limoges
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Metz-Tessy
  - GSK Investigational Site, Montauban
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Mûrs-Erigné
  - GSK Investigational Site, Nancy
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Narbonne
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Obernai
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Perpignan
  - GSK Investigational Site, Rosiers-d'Égletons
  - GSK Investigational Site, Rouen
  - GSK Investigational Site, Royaumeix
  - GSK Investigational Site, Saint-Etienne
  - GSK Investigational Site, Saint-Ouen-la-Rouërie
  - GSK Investigational Site, Scorbé-Clairvaux
  - GSK Investigational Site, Segré
  - GSK Investigational Site, Soulac-sur-Mer
  - GSK Investigational Site, Strasbourg
  - GSK Investigational Site, Thouars
  - GSK Investigational Site, Toul
  - GSK Investigational Site, Toulon
  - GSK Investigational Site, Toulouse
  - GSK Investigational Site, Verzy
  - GSK Investigational Site, Vieux-Condé
  - GSK Investigational Site, Villejuif
  - GSK Investigational Site, Wattrelos
  - GSK Investigational Site, Witry-lès-Reims
- Germany (13):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Wallerfing, Bavaria
  - GSK Investigational Site, Potsdam, Brandenburg
  - GSK Investigational Site, Dortmund, North Rhine-Westphalia
  - GSK Investigational Site, Rheine, North Rhine-Westphalia
  - GSK Investigational Site, Delitzsch, Saxony
  - GSK Investigational Site, Leipzg, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Teuchern, Saxony-Anhalt
  - GSK Investigational Site, Geesthacht, Schleswig-Holstein
  - GSK Investigational Site, Schmölln, Thuringia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Magdeburg

REFERENCES:
- [Derived] Devillier P, Humbert M, Boye A, Zachgo W, Jacques L, Nunn C, West S, Nicholls A, Antoun Z, Spinu L, Grouin JM. Efficacy and safety of once-daily fluticasone furoate/vilanterol (FF/VI) versus twice-daily inhaled corticosteroids/long-acting beta2-agonists (ICS/LABA) in patients with uncontrolled asthma: An open-label, randomized, controlled trial. Respir Med. 2018 Aug;141:111-120. doi: 10.1016/j.rmed.2018.06.009. Epub 2018 Jun 9. PMID 30053956

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 439 participants with persistent asthma were screened. The study was conducted at 63 centers in 2 countries: 43 in France and 20 in Germany from 09 July 2015 to 20 July 2017. Age value being reported for all participants is an approximate age accurate to within + or -1 year.
Pre-assignment Details: A total of 439 participants were screened for this study and 423 participants were randomized to treatment. Three of the randomized participants did not receive study treatment and were not included in the Intent-To-Treat (ITT) population.
Groups:
- Usual ICS/LABA: Eligible participants received fixed combination inhaled corticosteroid (ICS)/long-acting beta2-agonist (LABA) (Fluticasone propionate [FP]/ Salmeterol [S] 250/50 micrograms [mcg] or 500/50 mcg, 1 inhalation twice daily; or Budesonide [BUD]/ Formoterol [F] 200/6 mcg or 400/12 mcg, 1 or 2 inhalations twice daily) for 24 weeks.
- FF/VI: Eligible participants received Fluticasone Furoate (FF)/ Vilanterol (VI) 100 mcg/22 mcg or FF/VI 200 mcg/25 mcg 1 inhalation once daily for 24 weeks.
Period: Overall Study
Arm/Group | Usual ICS/LABA | FF/VI
Started | 210 | 210
Completed | 192 | 194
Not Completed | 18 | 16
Not completed — Adverse Event | 4 | 8
Not completed — Physician Decision | 5 | 1
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Lost to Follow-up | 2 | 2
Not completed — Protocol Violation | 1 | 2
Not completed — Lack of Efficacy | 2 | 0
Not completed — Protocol defined stopping criteria reach | 1 | 0

BASELINE CHARACTERISTICS:
Population: ITT Population comprised of all randomized participants who received at least one dose of the prescription of study medication (either FF/VI or usual ICS/LABA).
Groups:
- Usual ICS/LABA: Eligible participants received fixed combination ICS/LABA (FP/S 250/50 mcg or 500/50 mcg, 1 inhalation twice daily; or BUD/F 200/6 mcg or 400/12 mcg, 1 or 2 inhalations twice daily) for 24 weeks.
- FF/VI: Eligible participants received Fluticasone FF/Vilanterol VI 100 mcg/22 mcg or FF/VI 200 mcg/25 mcg 1 inhalation once daily for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Usual ICS/LABA | FF/VI | Total
Number analyzed (Participants) | 210 | 210 | 420
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.5 (14.99) | 49.3 (14.67) | 48.4 (14.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 145 | 269
  Male | 86 | 65 | 151
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 3 | 4 | 7
  Asian - Central/South Asian Heritage | 0 | 1 | 1
  Asian - East Asian Heritage | 2 | 0 | 2
  Asian - South East Asian Heritage | 0 | 1 | 1
  Native Hawaiian Or Other Pacific Islander | 1 | 1 | 2
  White - Arabic/North African Heritage | 8 | 6 | 14
  White - White/Caucasian/European Heritage | 196 | 196 | 392
  Mixed White Race | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Asthma Control Test (ACT) Total Score at Week 12
Description: The ACT is a validated self-completed questionnaire consisting of 5 questions that evaluate asthma control during the past 4 weeks on a 5-point categorical scale. Total scores are calculated from the sum of the scores from the 5 questions and can range from 5 to 25, with higher scores indicating better control. An ACT total score of 5 to 19 suggests that the participant's asthma is unlikely to be well controlled, whilst a score of 20 to 25 suggests that the participant's asthma is likely to be well controlled. Baseline value was the last assessment prior to randomization (Day 0). Change from Baseline was post-dose visit value minus the Baseline value. Least square mean change is presented.
Time Frame: Baseline and Week 12
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Usual ICS/LABA | FF/VI
Number analyzed (Participants) | 188 | 188
Scores on a Scale | 2.8 (0.26) | 3.6 (0.26)
Statistical Analysis 1: Comparison: Usual ICS/LABA vs FF/VI; Test type: Non-Inferiority — Non-inferiority of fixed combination FF/VI to usual ICS/LABA in inhalation powder was assessed assuming a non-inferiority margin of -1.5; p = 0.033, Mixed model repeated measures (MMRM); Mean Difference (Net) = 0.8, 95% CI 2-sided [0.1 to 1.5]; The analysis method was an MMRM adjusted for randomized treatment, visit (Week 6 and Week 12), Baseline ACT total score, randomized treatment-by-visit interaction, Baseline ACT total score-by-visit interaction, gender, age, country and participant fitted as a random factor. The Restricted Maximum Likelihood (REML) estimation approach was used with a default covariance structure of unstructured

2. Secondary Outcome: Change From Baseline in ACT Total Score at Week 24
Description: The ACT is a validated self-completed questionnaire consisting of 5 questions that evaluate asthma control on a 5-point categorical scale. Total scores are calculated from the sum of the scores from the 5 questions and can range from 5 to 25, with higher scores indicating better control. An ACT total score of 5 to 19 suggests that the participant's asthma is unlikely to be well controlled, whilst a score of 20 to 25 suggests that the participant's asthma is likely to be well controlled. Baseline value was the last assessment prior to randomization (Day 0). Change from Baseline was post-dose visit value minus the Baseline value. Least square mean change is presented.
Time Frame: Baseline and Week 24
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Usual ICS/LABA | FF/VI
Number analyzed (Participants) | 184 | 180
Scores on a Scale | 3.6 (0.25) | 4.0 (0.25)
Statistical Analysis 1: Comparison: Usual ICS/LABA vs FF/VI; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.224, Mixed model repeated measures (MMRM); Mean Difference (Net) = 0.4, 95% CI 2-sided [-0.3 to 1.1]; The analysis method was an MMRM adjusted for randomized treatment, visit (Week 6, Week 12, Week 18 and Week 24), Baseline ACT total score, randomized treatment-by-visit interaction, Baseline ACT total score-by visit interaction, gender, age, country and participant fitted as a random factor. The REML estimation approach was used with a default covariance structure of unstructured

3. Secondary Outcome: Percentage of Participants With Correct Use of Device, Defined as Not Making Any Critical or Non-critical Errors, at Week 12, and at Week 24 Independently of the Use at Week 12
Description: Participants were asked to read the appropriate package insert for their prescribed inhaler and then the investigator (or suitably qualified designee) demonstrated the proper use of the inhaler. The participant was then asked to self-administer their first dose of study treatment under the supervision of the investigator and any critical and non-critical errors were recorded. Individual instruments for assessing correct inhaler use were provided for each of the three devices used in this study.
Time Frame: Week 12 and Week 24
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Usual ICS/LABA | FF/VI
Number analyzed (Participants) | 210 | 210
Percentage of participants
  Week 12; n= 195, 197: number analyzed (Participants) | 195 | 197
  Week 12; n= 195, 197 | 93 | 94
  Week 24; n= 191, 192: number analyzed (Participants) | 191 | 192
  Week 24; n= 191, 192 | 96 | 97
Statistical Analysis 1: Comparison: Usual ICS/LABA vs FF/VI; Week 12; Test type: Superiority; p = 0.820, Regression, Logistic; Adjusted Odds Ratio = 1.11, 95% CI 2-sided [0.47 to 2.62]; The analysis method was logistic regression adjusted for randomized treatment, correct use of inhaler device at Baseline, gender, age and country
Statistical Analysis 2: Comparison: Usual ICS/LABA vs FF/VI; Week 24; Test type: Superiority; p = 0.566, Regression, Logistic; Adjusted Odds Ratio = 1.41, 95% CI 2-sided [0.43 to 4.60]; [other analysis details as in outcome 3, analysis 1]

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse drug reactions were collected from start of study treatment up to Week 24
Description: On-treatment SAEs and non-serious adverse drug reactions were collected for the Safety Population comprised of all enrolled participants who received at least one dose of study medication (either FF/VI or usual ICS/LABA) and considered as-treated.
Arm/Group | Usual ICS/LABA | FF/VI
All-Cause Mortality (participants affected / at risk) | 0/210 | 0/209
Serious Adverse Events (participants affected / at risk) | 4/210 | 3/209
Other Adverse Events (participants affected / at risk) | 0/210 | 0/209
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual ICS/LABA (N=210) | FF/VI (N=209)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Labyrinthitis (Infections and infestations) | 0 (0) | 1 (1)
Ovarian abscess (Infections and infestations) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Adnexa uteri pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Varicose vein ruptured (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-04-28): https://cdn.clinicaltrials.gov/large-docs/18/NCT02446418/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-21): https://cdn.clinicaltrials.gov/large-docs/18/NCT02446418/SAP_001.pdf